CLINICAL TRIAL: NCT03253289
Title: A Window of Opportunity Trial with Meclizine in Hepatocellular Carcinoma
Brief Title: Meclizine for Hepatocellular Carcinoma
Acronym: OPTIM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tannaz Armaghnay (Other)
Responsible Party: Sponsor-Investigator, Tannaz Armaghnay, Assistant Professor of Medicine - Hematology and Oncology, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-40370
Record Dates: First submitted 2017-05-19; First posted 2017-08-17 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Hepatocellular carcinoma, HCC, Liver cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Meclizine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Meclizine 100 mg (Experimental): Meclizine 50 mg will be taken by the patient orally twice daily for a total of 28 days(up to 35 days).
  Interventions: Drug: Meclizine Oral Tablet

INTERVENTIONS:
Drug: Meclizine Oral Tablet — All subjects will receive 50 mg of meclizine taken orally, twice a day (daily dose 100 mg) for 28 (up to 35) days.

SUMMARY:
Meclizine hydrochloride is an antihistamine widely used for treatment of vertigo and motion sickness. In HCC it has been used for anti-emetic effects, but it is used here as a CAR (constitutive androstane receptor) inverse agonist.

The hypothesis of this study is that Meclizine, CAR inverse agonist, will have beneficial therapeutic effect in patients with hepatocellular carcinoma who are candidates for surgical resection, ablation, TACE, Y90 or systemic therapy by blocking tumorigenesis and inducing apoptosis. The effects of Meclizine will be analyzed by measuring messenger RNA level of CAR target genes CYP2B6, c-Myc and FoxM1, the downstream effectors of CAR, by real time quantitative PCR.

DETAILED DESCRIPTION:
The constitutive androstane receptor (CAR, NR1I3) is a nuclear receptor that plays a central role in hepatic detoxification of potentially toxic compounds, or xenobiotics. Chronic CAR activation by specific agonists induces tumors in wild type mice, and strongly promotes hepatocarcinogenesis in combination with initiating mutagens. Both effects are absent in CAR null mice. These tumorigenic effects are associated with an acute induction of hepatocyte proliferation in mice. Preliminary results using partially humanized mice demonstrate a very similar proliferative effect of CAR activation in human hepatocytes.

The transcriptional activity of CAR can be reversed by specific inverse agonists. These ligands are analogous to steroid receptor antagonists, converting the transcriptional activation of the agonist bound receptor into transcriptional repression. These compounds are termed inverse agonists because they do not depend on the presence of agonist ligands to exert their repressive effects. Mouse and human CAR proteins are more divergent than other nuclear receptors, and respond to quite different profiles of agonists and inverse agonists. Preliminary results demonstrate that the specific mouse CAR inverse agonist androstanol blocks proliferation and induces apoptosis in mouse liver tumors. This raises the possibility that targeting CAR may represent a new modality of treatment for hepatocellular cancer (HCC) analogous to estrogen and androgen receptor antagonists in breast and prostate cancers. Meclizine, a widely used antihistamine medication for vertigo and motion sickness, is an inverse agonist ligand of human CAR. Investigators hypothesize that reversing CAR function with meclizine will have a beneficial therapeutic effect in patients with HCC by blocking proliferation and inducing apoptosis.

Investigators therefore propose a novel window of opportunity trial in which biopsy proven HCC patients will receive oral meclizine daily for 28 (up to 35) days while awaiting surgical resection, radiofrequency ablation, transarterial chemoembolization, Y90 or systemic therapy. The primary test of treatment outcome will be the predicted decrease in expression of downstream CAR target genes (CYP2B6, MYC and FOXM1) in pre and post treatment tumor specimens. Investigators will also measure the change in tumor proliferation and apoptosis by measuring Ki-67 proliferation index and TUNEL assays (terminal deoxynucleotidyl transferase dUTP Nick-End Labeling assay), serum levels of AFP and GDF 15, and overall tumor response by imaging. HCC is the most rapidly increasing cause of cancer mortality in the United States and medical treatment options are limited. Successful completion of this study may identify a new approach to treatment of HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have imaging: CT or MRI abdomen with and without contrast confirmed or highly suspicious for Hepatocellular carcinoma. Patients must have a liver biopsy confirmed for Hepatocellular carcinoma.
2. Patients must have measurable disease, defined as tumor mass which is >10 mm with spiral CT scan or MRI. Baseline imaging scan must be within 8 weeks of registration.
3. Patients must have no prior history of treatment for HCC (treatment naïve) on the lesion that is being targeted for biopsy. New HCC lesions can arise in the liver of patients despite local therapy of other areas of the liver due to consistent underlying risk factors such as cirrhosis, and chronic hepatitis B or C infection. Patients with prior local liver directed therapy such as TACE, Ablation, Y-90 or hepatectomy surgery for HCC are eligible if they have developed a new untreated lesion in the liver which can be targeted for a biopsy for this study. There is no required time frame or washout period from when a lesion has been locally treated to the time when a new lesion is found and targeted for biopsy for this trial. Patients who have had prior systemic therapy of any kind are not eligible.
4. Patients must be greater than 18 years of age.
5. ECOG Performance status less than/equal to 2 (Karnofsky greater than 60%).
6. Patients must have normal organ and marrow function as defined below, within 21 days of registration: Leukocytes greater than 3,000/mcL; ANC greater than 1,500/mcL; Platelets greater than 50,000/mcL; Hemoglobin greater than/equal to 8 g/dL; ALT(SGPT) less than/equal to 5X IULN and AST (SGOT) less than/equal to 5X IULN; Creatinine less than/equal to 2X IULN or Creatinine clearance greater than 60 mL/min for patients with creatinine levels greater than IULN; Child Pugh Class A (5-6 points) or B (7 points); INR less than/equal to 2.3; Albumin greater than 2.8 g/dL; Total bilirubin less than/equal to 3X IULN.
7. Patients must be candidate for surgical resection, ablation, TACE, Y90 or systemic therapy.
8. Patients should have life expectancy greater than/equal to 10 weeks.
9. Willingness to Use Contraception: The effects of Meclizine on the developing human fetus at the recommended therapeutic dose are unknown. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study treatment with meclizine. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. If a male participant impregnates his partner he should inform his treating physician immediately.
10. Patients must be informed of the investigational nature of this study, and must sign and give written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

1. Patients may not be receiving any other concurrent anti-cancer therapy.
2. Patients may not be receiving any other concurrent investigational agents.
3. Patients taking medications with a narrow therapeutic index including warfarin, digoxin, phenobarbital, carbamazepine, and cyclosporine are not excluded but should be monitored carefully.
4. Patients must not be taking Rifampin or St John's Wort.
5. Patient must not have a history of allergic reactions like anaphylaxis attributed to compounds of similar chemical or biologic composition to Meclizine such as antihistamine drugs.
6. Patient must not be a candidate for liver transplant.
7. Child Pugh Class B (8,9) and Class C are excluded
8. Antiviral therapy for HCV and HBV is allowed, but patient should not be on interferon.
9. HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with meclizine.
10. Patient must not have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction or cerebrovascular accident within 6 months prior to registration, cardiac arrhythmia, glaucoma, asthma or psychiatric illness/social situations that would limit compliance with study requirements.
11. Pregnant women are excluded from this study because meclizine is a Class B agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with meclizine, breastfeeding should be discontinued if the mother is treated with meclizine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Change in mRNA levels | day1 and last day of treatment(last day would be one time point between day 28 and day 35 of treatment)
  Quantitative real time PCR(qPCR) can give change in expression level compared to control Delta CT value. Downstream target genes of CAR (CYP2b6,c-Myc, and FoxM) will be measured by qPCR in the pre and post treatment Hepatocellular cancer tissue specimens. The qPCR machine measures the intensity of fluorescence emitted by the probe at each cycle. The Ct measure is a determined PCR cycle and represents the basic result of a qPCR experience. The Ct is the value where the PCR curve crosses the threshold.

SECONDARY OUTCOMES:
Change in Ki-67 proliferation index | day1 and last day of treatment(last day would be one time point between day 28 and day 35 of treatment)
  The proliferative index is a measure of the number of cells in a tumor that are dividing (proliferating).
change in apoptosis by TUNEL assay | day1 and last day of treatment(last day would be one time point between day 28 and day 35 of treatment)
  apoptosis will be measured by TUNEL (terminal deoxynucleotidyl transferase dUTP Nick-End Labeling assay)
Tumor response | day1 and last day of treatment(last day would be one time point between day 28 and day 35 of treatment)
  Assess tumor response by RECIST criteria
Change in Serum AFP | day1 and last day of treatment(last day would be one time point between day 28 and day 35 of treatment)
  This will be measured in peripheral blood samples
Change in growth differentiation factor (GDF-15) | day1 and last day of treatment(last day would be one time point between day 28 and day 35 of treatment)
  This will be measured in peripheral blood samples
A panel of CAR downstream target genes | day1 and last day of treatment(last day would be one time point between day 28 and day 35 of treatment)
  expression of a panel of CAR downstream target genes

CONTACTS AND LOCATIONS:
Overall Officials: Tannaz Armaghany, MD, Principal Investigator — Baylor College of Medicine
Locations (5):
- United States (5):
  - Baylor College of Medicine -McNair Campus, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Baylor St. Luke's Medical Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Harris Health System- Smith Clinic, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared, as indicated above.